CLINICAL TRIAL: NCT00565019
Title: The Effects of Steroid Injection With Percutaneous Needle Aponeurotomy in Patients With Dupuytren's Contracture: a Randomized Controlled Study
Brief Title: Effects of Steroid Injection With Percutaneous Needle Aponeurotomy in Dupuytren's Contracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Society of Plastic Surgeons (Other)
Responsible Party: Principal Investigator, Dr. Paul Binhammer, MD, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUPTRNS_STRD_RCT
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Steroid (Experimental)
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — * Triamcinolone acetonide will be administered into the cord following surgery with a tuberculin syringe and a 25-gauge needle.
  * Doses will range from 60-120 mg depending on extent of the disease.
  * Patients will receive injections at 6 weeks and 3 months for persisting nodules or cords.
  * PI will determine the dosages. Estimates will be made based on the following:
  Size of nodule/cord: 1-2 cm2, dosage 20-40 mg
  Size of nodule/cord: 2-6 cm2, dosage 40-80 mg
  Size of nodule/cord: 6-10 cm2, dosage 80-100 mg
  Size of nodule/cord: >10 cm2, dosage 100-120 mg
  Arms: Steroid

SUMMARY:
Background:

Dupuytren's contracture is a common hand problem that causes certain fingers to bend towards the palm. Patients with this condition cannot perform daily activities and many are unable to work. It is usually treated by an operation to straighten the fingers followed by therapy if the angle that the fingers are bent at is large enough. However, no treatment has been able to completely prevent the angle from persisting.

Objective:

This study is designed to examine whether or not the use of a drug in combination with surgery will improve the angle at which the fingers are bent more than surgery alone.

Hypothesis:

Subjects who receive triamcinolone acetonide will have straighter fingers compared with subjects who only have the operation and no triamcinolone acetonide at both 3 months and 6 months after the operation.

Methods:

Eligible patients interested in having the operation to treat Dupuytren's contracture will be asked if they would like to join the study. Subjects will be randomly placed into one of two groups: the steroid injection group or the control group. Subjects will have a pre-operative visit, the surgery, and follow-ups at 6 weeks, 3 months and 6 months. All subjects will have the operation, but only those in the steroid injection group will receive an injection of the drug. During the 6 week and 3 month follow-ups, subjects in the steroid injection group may receive another injection if their fingers are still bent. Angles are measured at the pre-operative visit and at 3 and 6 months. The change in angle from before to after and any differences in the groups, in time points and interactions between the two will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18.
* Literate in the English language.
* Diagnosed by the PI with Dupuytren's contracture with an angle of contracture of 20° or greater.
* Candidates for percutaneous needle aponeurotomy.
* First surgery on the affected digit.

Exclusion Criteria:

* Allergy or sensitivity to triamcinolone acetonide or any of the non-medicinal components in the suspension.
* Patient is not a candidate for steroid injection for other medical reasons, which will be determined by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the angle of contracture of the affected fingers (how bent the fingers are before and after the two treatments). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Binhammer, MD,MSc, Principal Investigator — Division of Plastic Surgery, Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Division of Plastic Surgery, Toronto, Ontario, Canada